CLINICAL TRIAL: NCT07016217
Title: Impact Evaluation of the Therapeutics Initiative's Mailed Dental Portrait and Therapeutics Letter
Brief Title: Evaluation of an Educational Intervention on Antibiotics in Dental Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government); British Columbia Centre for Disease Control (Other Government); British Columbia College of Oral Health Professionals (Unknown)
Responsible Party: Principal Investigator, Colin Dormuth, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: H23-01507
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Dental Infection; Clindamycin; Antibiotics
Keywords: randomized controlled trial; dental infection; clindamycin; quality improvement; prescribing feedback; antibiotics

STUDY DESIGN:
Intervention Model Description: The investigators randomized actively practicing dentists into three groups, n=1166 in each group for a total of 3498 individual dentists.
  For the Early mailing on Oct 13, 2023, Arm A/Group 1 received the "plain" Portrait with a Therapeutics Letter; Arm B/Group 2 received a "complete" Portrait with a Letter, and Arm C/ Group 3 received nothing (control group). For the delayed mailing (April 24, 2024), Arm A/Group 1 received the "complete" Portrait and Letter, Arm B/Group 2 received nothing, and Arm C/ Group 3 received the "plain" Portrait and Letter.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Group 1) - Portrait + Letter (Experimental): This group received the "plain" Portrait with a Therapeutics Letter in the Early mailing (Oct 13, 2023), and received the "complete" Portrait with a Therapeutics Letter in the Delayed mailing (April 24, 2024).
  Interventions: Behavioral: Early Plain Portrait and Letter; Behavioral: Delayed Complete Portrait
- Arm B (Group 2) - Portrait + Letter (Experimental): This group received the "complete" Portrait with a Therapeutics Letter in the Early mailing (Oct 13, 2023), and received nothing in the Delayed mailing (April 24, 2024).
  Interventions: Behavioral: Early Complete Portrait and Letter; Behavioral: No intervention
- Arm C (Group 3) - Control (Experimental): This group received nothing in the Early mailing (Oct 13, 2023) and received the "plain" Portrait with a Therapeutics Letter in the Delayed mailing (April 24, 2024).
  Interventions: Behavioral: No intervention; Behavioral: Delayed Plain Portrait and Letter

INTERVENTIONS:
Behavioral: Early Plain Portrait and Letter — In the context of audit and feedback interventions, the prescribing Portrait is a document produced by the Therapeutics Initiative that provides personalized prescribing feedback for clinicians in British Columbia. Portraits are used as a practice resource tool for reflection on prescribing or test-ordering patterns.
  The Portraits provide data of individual prescribing along with evidence-based benchmarks or targets. The "plain" Portrait includes the main message, prescriber's data (compare to optimal prescribing, with or without information on BC mean/median). Prescribers are also given access to a succinct review of the best available evidence on the topic and recommendations for future action in the Therapeutics Letter, a standalone publication that details the evidence for the recommended practice in a brief and practical manner, with references.
  Arms: Arm A (Group 1) - Portrait + Letter
Behavioral: Early Complete Portrait and Letter — In the context of audit and feedback interventions, the prescribing Portrait is a document produced by the Therapeutics Initiative that provides personalized prescribing feedback for clinicians in British Columbia. Portraits are used as a practice resource tool for reflection on prescribing or test-ordering patterns.
  The Portraits provide data of individual prescribing along with evidence-based benchmarks or targets. The "complete" Portrait includes the main message, prescriber's data (compare to optimal prescribing, with or without information on BC mean/median) and a series of self-reflection questions. Prescribers are also given access to a succinct review of the best available evidence on the topic and recommendations for future action in the Therapeutics Letter, a standalone publication that details the evidence for the recommended practice in a brief and practical manner, with references.
  Arms: Arm B (Group 2) - Portrait + Letter
Behavioral: No intervention — To measure the impact of the interventions, Arm C (Group 3) will receive no intervention in the Early mailing and Arm B (Group 2) will receive no intervention in the Delayed mailing.
  Arms: Arm B (Group 2) - Portrait + Letter; Arm C (Group 3) - Control
Behavioral: Delayed Plain Portrait and Letter — Delayed "plain" Portrait and Letter (as described)
  Arms: Arm C (Group 3) - Control
Behavioral: Delayed Complete Portrait — Delayed "complete" Portrait and Letter (as described)
  Arms: Arm A (Group 1) - Portrait + Letter

SUMMARY:
The goal of this randomized trial is to estimate the impact of personalized prescribing portraits and educational materials on prescribing of antibiotic medications by dentists in British Columbia, Canada.

The main research question is:

Did the prescribing Portraits and Therapeutics Letter lead to a change in clindamycin prescribing as a proportion of total antibiotic prescribing by dentists in British Columbia.

Study participants are dentists actively practicing in British Columbia. Participants were randomized to 3 study arms to received different combinations of one of two versions of the individual prescribing Portraits and a Therapeutics Letter in Early or Delayed Groups. Two versions of the prescribing Portrait were used: a "plain" version and a "complete" version, which included an additional section with self-reflection questions for clinicians.

Using administrative health data, the prescribing of those in different combinations of materials in the Early Group will be compared to those in the Delayed Group to estimate the impact of the materials on prescribing by the dentists.

DETAILED DESCRIPTION:
Audit and feedback is a well-established strategy for improving the quality of care in primary healthcare settings. It involves the systematic collection and analysis of healthcare data, followed by the provision of information to healthcare providers to improve the quality of care.

Based in British Columbia, Canada, the Therapeutics Initiative's Portrait program provides physicians, and other health professionals, with individualized prescribing data compared with their peers, paired with evidence-based messaging, and a concise statement summarizing the desired change in prescribing behavior. The Portrait program implements a series of pragmatic trials to improve prescribing where clinicians are randomized into an early intervention and a delayed control group.

This study is a randomized trial examining the impact of prescribing Portraits on antibiotic prescribing by dentists in British Columbia. The Portrait title is "Which antibiotics do you prescribe for dental infections?" and is accompanied by a Therapeutics Letter entitled "Rethink Clindamycin for Dental Patient Safety." The materials were developed in collaboration with the BC Centre for Disease Control (BCCDC) and the BC College of Oral Health Professionals (BCCOHP).

When dentists prescribe antibiotics like clindamycin for dental infections, they often do so with the intention of combating bacterial growth. However, clindamycin come with a set of risks, notably the potential for Clostridium difficile infection (C. diff). This bacterium can proliferate in the gut when the normal balance of bacteria is disrupted by antibiotics, leading to symptoms ranging from mild diarrhea to severe colitis and life-threatening complications.

The main prescribing message for the dental Portrait is "clindamycin should not be used routinely for prophylaxis or management of dental infections." The Portrait has two different formats. The "plain" version includes the main message, prescriber's data (compare to optimal prescribing), and references. The "complete" version includes an additional series of self-reflection questions.

3498 dentists in British Columbia were randomized into three arms/groups (1166 in each group). For the Early mailing in Oct 2023, Arm A received the "plain" Portrait with a Therapeutics Letter; Arm B received a "complete" Portrait with a Letter, and Arm C received nothing. For the delayed mailing (April 2024), Arm A received the "complete" Portrait and Letter, Arm B received nothing, and Arm C received the "plain" Portrait and Letter.

The objective was to estimate the impact of the interventions (plain version of Portrait + Therapeutics Letter; Complete version of the Portrait + Therapeutics Letter; repeat messages) on prescribing of antibiotic medications by dentists in British Columbia.

The analysis will identify:

* Baseline characteristics: Physicians and patients by study group (age, age groups, and sex).
* Primary outcome: The change in clindamycin prescribing as a proportion of total antibiotic prescribing associated with the Portraits and Therapeutics Letter.

The investigators will identify the difference in the number of new starts of clindamycin after versus before the Early mailing date. New starters of clindamycin are defined as no antibiotic prescribed by any dentist in the previous year. Investigators will then calculate the mean difference among dentists in each of the comparison groups by estimating the odds ratio: adjust for clustering using GEE, with an interaction term between the randomization group id and time period, and with an independent correlation structure. Analysis assumes a normal distribution to derive confidence intervals. The difference between the comparison groups will be the estimated impact of the portrait.

Analysis will be conducted using secondary data from administrative databases from the BC Ministry of Health (under an Information Sharing Agreement). The data are patient level and include anonymized information about demographics, health costs, BC Medical Services Plan clinician services data, BC PharmaNet data (prescription drug dispensing at community pharmacies), client roster. The data do not include personally identifiable patient information.

ELIGIBILITY:
Inclusion Criteria:

* Dentists registered with the BC College of Oral Health Professionals with an active dental practice in BC
* Dentists in BC included in randomization groups 1-3 with at least 10 prescription orders filled for antibiotics in 2022
* Patients aged >16
* Patient prescribed antibiotic therapy by a BC dentist during, before, or after periods; Anatomical Therapeutic Chemical (ATC) classes J01
* Patient was enrolled in MSP at least 1 month before the prescription

Exclusion Criteria:

* Dentists not registered with the BC College of Oral Health Professionals
* Dentists with fewer than 10 prescription orders filled in 2022
* Patients used antibiotics in the last 14 days (prescribed by any prescriber, not only dentists) before the prescription; and
* Federally insured BC residents and beneficiaries of the First Nations Health Benefit Plan; we were not given permission to use these data in our evaluation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3498 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Intention to treat analysis | Assessed from the baseline until the early intervention (6 months) to 6 months after the delayed intervention (total of 18 months).
  The primary outcome is the change in clindamycin prescribing (number of new starts) as a proportion of total antibiotic prescribing associated with the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, ScD, Principal Investigator — University of British Columbia
Locations (1):
- Therapeutics Initiative - Dept of Anesthesiology, Pharmacology & Therapeutics, Faculty of Medicine, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The data access agreement for the Therapeutics Initiative does not permit sharing of IPD.